CLINICAL TRIAL: NCT07404956
Title: COMPARISON OF THE EFFECTS OF SURGICAL MASK AND N95 MASK USE ON PHYSICAL SYMPTOMS OF SURGICAL SMOKE IN OPERATING ROOM
Brief Title: THE EFFECT OF SURGICAL MASK AND N95 MASK USE ON SURGICAL SMOKE IN OPERATING ROOM NURSES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Hilal Çetin Baltutar, Nurse, Bartın Unıversity
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BARU-SBF-2025-01
Record Dates: First submitted 2025-12-31; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Surgical Smoke Exposure; Occupational Exposure to Surgical Smoke; Headache; Dizziness; Nause and Vomiting; Fatigue Symptom; Eye Allergies; Abdominal Pain (AP); Heart Rate Determination; SpO2; Muscle Weakness | Patient; Muscle Aches; Dispnea
Keywords: Surgical Smoke; Masks; Operating Room Nurses; Occupational Exposure
MeSH Terms: conditions — Headache; Dizziness; Vomiting; Fatigue; Abdominal Pain; Myalgia | interventions — N95 Respirators

STUDY DESIGN:
Masking Description: Outcome assessment and data analysis were conducted by an independent assessor blinded to the type of mask used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Mask (Experimental): Operating room nurses used a standard surgical mask during surgical procedures with exposure to surgical smoke.
  Interventions: Device: Surgical Mask
- N95 Mask (Experimental): Operating room nurses used an N95 respirator during surgical procedures with exposure to surgical smoke.
  Interventions: Device: N95 Mask

INTERVENTIONS:
Device: Surgical Mask — Standard surgical masks were used by operating room nurses during surgical procedures with exposure to surgical smoke.
  Other Names: Medical Surgical Mask
  Arms: Surgical Mask
Device: N95 Mask — N95 respirators were used by operating room nurses during surgical procedures with exposure to surgical smoke.
  Other Names: N95 Respirator
  Arms: N95 Mask

SUMMARY:
This study was conducted to compare the effect of surgical mask and N95 mask use on physical symptoms due to surgical smoke in operating theatre nurses. The study, which was conducted in a single-group prospective quasi-experimental design, was completed with 38 nurses in the operating theatre unit of a state hospital in the Western Black Sea Region. Data were collected for four weeks using the Descriptive Information Form, Numerical Rating Scale and Symptom Follow-up Form. According to the findings, muscle weakness, myalgia in the upper extremities and muscle cramps were statistically significantly less in nurses using N95 masks. Respiratory parameters, watery eyes and redness were significantly lower in nurses using surgical masks. As a result, it was determined that the type of mask was effective on the incidence of physical symptoms related to surgical smoke.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Aged 18 years or older
* Working as a sterile operating room nurse at least 4 hours per day, 5 days per week
* Compliance with the protocol requiring continuous use of both surgical mask and N95 mask for at least 4 hours per day
* Ability to communicate verbally and provide informed consent

Exclusion Criteria:

* Diagnosed psychiatric disorders
* Presence of chronic respiratory, musculoskeletal, or neurological diseases
* Presence of chronic dermatological conditions or allergies affecting the facial or respiratory area
* Speech or communication impairments
* Pregnancy
* Holding a supervisory role (e.g., charge nurse) or non-sterile nursing role
* Planned unit change or rotation during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Surgical Smoke-Related Physical Symptom Severity (Total NRS Score) | Five days per week for a duration of four weeks both preoperatively and postoperatively
  The severity of physical symptoms related to surgical smoke exposure in operating room nurses, including headache, abdominal pain, nausea and vomiting, fatigue/weakness, loss of appetite, and dyspnea, was assessed using the Numeric Rating Scale (NRS). Each symptom was rated on a standardized numeric scale, and a total symptom severity score was calculated by summing the individual symptom scores. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: sevim çelik, Professor, Principal Investigator — Bartin University Health Science Faculty
Locations (1):
- Bartın State Hospital, Bartın, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No